CLINICAL TRIAL: NCT02312414
Title: Effects of Carnitine on Oxidative Stress and Inflammatory Responses to Intravenous Iron Administration to Patients With CKD: Impact of Haptoglobin Genotype
Brief Title: Effects of Carnitine on Oxidative Stress to IVIR Administration to CKD Patients:Impact of Haptoglobin Genotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Nazareth Hospital, Israel (Other)
Responsible Party: Principal Investigator, zaher armaly, Dr Zaher Armaly, Head of Nephrology and Hypertension Department Nazareth Hospital- EMMS, Nazareth Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5700858
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIR (No Intervention): Patients given IV iron (Sodium ferric gluconate, [125 mg/100 ml] from week 1 to week 4
- IVIR Carnitine (Experimental): Patients given Carnitine (20mg/kg, IV) perior to IV iron (Sodium ferric gluconate, [125 mg/100 ml] from week 4 to week 8.
  Interventions: Drug: L-Canitine

INTERVENTIONS:
Drug: L-Canitine — Carnitine is a quaternary ammonium compound biosynthesized from the amino acids lysine and methionine, it is essential for the transport of fatty acids from the intermembraneous space in the mitochondria, into the mitochondrial matrix during the breakdown of lipids (fats) for the generation of metabolic energy
  Arms: IVIR Carnitine

SUMMARY:
Anemia is a common disorder in CKD patients. It is largely attributed to decreased erythropoietin (EPO) production and iron deficiency. Therefore, besides EPO, therapy includes iron replenishment. However, the latter induces oxidative stress. Haptoglobin (Hp) protein is the main line of defense against the oxidative effects of Hemoglobin/Iron. There are 3 genotypes: 1-1, 2-1 and 2-2. Hp 2-2 protein is inferior to Hp 1-1 as antioxidant. So far, there is no evidence whether haptoglobin genotype affects iron-induced oxidative stress in CKD patients.

In this proposed study we wished to examine whether Hp genotype influences intravenous iron administration (IVIR)-induced oxidative stress in CKD patients, and its impact on the response of these patients to L-Carnitine therapy.

DETAILED DESCRIPTION:
This study will include at least 25 anemic CKD patients (stages 3-4) that will be given a weekly IVIR (Sodium ferric gluconate, [125 mg/100 ml] for 8 weeks, and during weeks 5-8 also received Carnitine (20mg/kg, IV) prior to IVIR. Weekly blood samples will drawn before and after each IVIR for Hp genotype, C-reactive protein (CRP), advanced oxidative protein products (AOPP), neutrophil gelatinase-associated lipocalin (NGAL), besides complete blood count and biochemical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have been diagnosed as suffering from chronic kidney diseases at stages 3-4 and confirmed by MDRD.
2. CKD patients with Hb of less than 10 g%.
3. At age ≥18 y.

Exclusion Criteria:

1. Pregnant women.
2. Patient with CKD stage 5 on Dialysis.
3. Patients with severe liver diseases.
4. Patients with severe CHF.
5. Inter-current illness such as fever.
6. Allergic rhinitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
AOPP (Advanced Oxidation Protein Products) | 1 month
neutrophil gelatinase-associated lipocalin (NGAL), | 1 month

SECONDARY OUTCOMES:
Haptoglobin | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Amir Abd El Qader, Ph.D, Study Director — Nazareth EMMS Hospital
Locations (1):
- Nazareth hospital (EMMS), Nazareth, Israel

REFERENCES:
- [Derived] Armaly Z, Abd El Qader A, Jabbour A, Hassan K, Ramadan R, Bowirrat A, Bisharat B. Effects of carnitine on oxidative stress response to intravenous iron administration to patients with CKD: impact of haptoglobin phenotype. BMC Nephrol. 2015 Aug 13;16:135. doi: 10.1186/s12882-015-0119-0. PMID 26268514